CLINICAL TRIAL: NCT02867657
Title: Enhancement of Presence, Compassion and Resilience Bringing the Practice of Mindfulness Into Nature - Preventing Mental Fatigue in Healthcare Professionals.
Brief Title: Bringing the Practice of Mindfulness Into Nature - Preventing Mental Fatigue in Healthcare Professionals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIA University College (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: H-15010925
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2018-02

CONDITIONS: Stress, Psychological; Inflammation; Stress, Physiological
MeSH Terms: conditions — Stress, Psychological; Inflammation | interventions — Mindfulness; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness in nature (Experimental): A five day mindfulness retreat in nature
  Interventions: Behavioral: Mindfulness
- Mindfulness indoor (Active Comparator): A five day mindfulness retreat indoor
  Interventions: Behavioral: Mindfulness
- Wait list control (No Intervention): A wait list control group, that 6 months later is offered a two-day mindfulness retreat in nature

INTERVENTIONS:
Behavioral: Mindfulness — Five days MBSR curriculum with meditation and yoga
  Other Names: Mindfulness Based Stress Reduction; MBSR
  Arms: Mindfulness in nature; Mindfulness indoor

SUMMARY:
The purpose of the study is to determine whether a five day mindfulness retreat in nature can increase measures of attention and self-compassion, and reduce stress among bachelor students at Danish Universities and University Colleges. Secondary whether the expression of inflammatory markers can be reduced .

It is the hypothesis that perceived stress is reduced and the expression of genetic markers of inflammation is reduced after a five day mindfulness retreat.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor student at a Danish University or University College
* A score of 16 or above on the Perceived Stress Scale (PSS)

Exclusion Criteria:

* Smoking
* Psychiatric diagnosis (depression, anxiety, adjustment disorder, PTSD, personality disorder, psychosis).
* Untreated ADHD, autism, abuse and risk of suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | At the end of five days retreat
  PSS
Self-compassion | At the end of five days retreat
  S-C-S Neff2

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire | At the end of five days retreat
Breath Counting | At the end of five days retreat
  Behavioral measurement of attention
NF-kB gene expression | At the end of five days retreat
IL-1 gene expression | At the end of five days retreat
IL-6 gene expression | At the end of five days retreat
cRP expression | At the end of five days retreat
  c reactive protein
Heart Rate Variability | At the end of five days retreat
  HRV
Blood pressure | At the end of five days retreat
Connectedness to Nature Scale | At the end of five days retreat
GR gene expression | At the end of five days retreat
RIPK2 gene expression | At the end of five days retreat
TNF-α gene expression | At the end of five days retreat
CCL5 gene expression | At the end of five days retreat
IL-8 gene expression | At the end of five days retreat
TERT gene expression | At the end of five days retreat
TERC gene expression | At the end of five days retreat
IL-1β protein expression | At the end of five days retreat
IL-2 protein expression | At the end of five days retreat
IL-4 protein expression | At the end of five days retreat
IL-6 protein expression | At the end of five days retreat
IL-8 protein expression | At the end of five days retreat
IL-10 protein expression | At the end of five days retreat
IL-12p70 protein expression | At the end of five days retreat
IL-13 protein expression | At the end of five days retreat
TNF-α protein expression | At the end of five days retreat
IFN-γ protein expression | At the end of five days retreat

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - VIA University College, Aarhus
  - Nacadia, University of Copenhagen, Hoersholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879